CLINICAL TRIAL: NCT04441242
Title: Use of Ambient Lighting During Colonoscopy and Its Effect on Adenoma Detection Rate and Eye Fatigue: a Pilot Study
Brief Title: Ambient Lighting During Colonoscopy and Its Effect on Adenoma Detection Rate and Eye Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 6665
Record Dates: First submitted 2020-06-02; First posted 2020-06-22 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Cancer Screening; Colon Adenomatous Polyp

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrospective: Low lighting during screening colonoscopy (Placebo Comparator): Screening colonoscopies performed with low lighting conditions.
  Interventions: Other: Low lighting
- Prospective: Ambient lighting during screening colonoscopy (Active Comparator): Screening colonoscopies performed with ambient lighting conditions.
  Interventions: Other: Ambient lighting

INTERVENTIONS:
Other: Ambient lighting — Use of ambient lighting (75-150 lux) in endoscopy room.
  Arms: Prospective: Ambient lighting during screening colonoscopy
Other: Low lighting — Use of low lighting (<75 lux) in endoscopy room.
  Arms: Retrospective: Low lighting during screening colonoscopy

SUMMARY:
A retrospective and prospective study to determine if the use of ambient lighting during screening colonoscopy is well tolerated and if ambient lighting will help physicians maintain adenoma detection rates while decreasing symptoms of eye strain as the day progresses.

DETAILED DESCRIPTION:
This study is a a single-center study at an independent community-based teaching hospital comparing adenoma detection rate in screening colonoscopies performed in low lighting with those performed with ambient lighting (75-150 lux). All cases included in the study involved adult patients undergoing screening colonoscopy with a participating gastroenterologist. Diagnostic colonoscopies, history of colon resection, colorectal cancer, and cases performed in children, pregnant women, and prisoners were excluded from analysis. Cases involving gastroenterology fellows were also excluded. Retrospective data was collected over a six month period from January 2017 to June 2017, followed by a prospective arm the during the same calendar months the subsequent year (January 2018 to June 2018).

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing screening colonoscopy
* Procedure performed by a participating gastroenterologist

Exclusion Criteria:

* Any diagnostic colonoscopies
* History of colon resection
* History of colorectal cancer
* Children
* Pregnant women
* Prisoners
* Cases involving trainees, including gastroenterology fellows

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1109 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in adenoma detection rate | 6 months
  Adenoma detection rate, comparing change from first case of the day to the last. Ranges from 0-99%, with greater increases adenoma detection rate (ADR) being more favorable.
Eye strain score | 6 months
  Eye strain score, as calculated from survey responses completed by physicians. Ranges from 0 - 60, with lower scores indicating less severe symptoms (therefore, lower scores are more favorable).

SECONDARY OUTCOMES:
Adenoma detection rate (overall) | Participants each assessed on one day during 6 month study period
  Overall adenoma detection rate. Ranges from 0% to 100%. Higher ADR is more favorable.
Adenoma detection rate (first case vs last case of the day) | Participants each assessed on one day during 6 month study period
  Adenoma detection rate, comparing first case of the day to the last. Ranges from from -99 to 99%, with greater numbers (increases) being more favorable.
Satisfaction by staff | 6 months
  Satisfaction by staff involved in endoscopy, based on survey responses

CONTACTS AND LOCATIONS:
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hayes JR, Sheedy JE, Stelmack JA, Heaney CA. Computer use, symptoms, and quality of life. Optom Vis Sci. 2007 Aug;84(8):738-44. doi: 10.1097/OPX.0b013e31812f7546. PMID 17700327
- [Result] Almadi MA, Sewitch M, Barkun AN, Martel M, Joseph L. Adenoma detection rates decline with increasing procedural hours in an endoscopist's workload. Can J Gastroenterol Hepatol. 2015 Aug-Sep;29(6):304-8. doi: 10.1155/2015/789038. Epub 2015 May 21. PMID 25996612